CLINICAL TRIAL: NCT06983301
Title: A Feasibility Study of Brief Cognitive Behaviour Therapy for Adolescent OCD in Routine Clinical Practice
Brief Title: Brief Cognitive Behaviour Therapy (CBT) for Adolescent OCD in Routine Clinical Practice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18475; 348693 (Other: IRAS Number)
Record Dates: First submitted 2025-04-01; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Obsessive Compulsive Disorder (OCD); CBT
Keywords: OCD; Adolescent mental health; CBT; Cognitive Behavioural Therapy; Brief psychological therapy; Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: This study is a multicentre single-arm (no blinding) feasibility intervention trial implementing brief CBT (supplemented with workbooks) to treat adolescents who meet diagnostic criteria for OCD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Brief CBT for OCD intervention delivered
  Interventions: Other: Brief Cognitive Behavioural Therapy (CBT) for OCD

INTERVENTIONS:
Other: Brief Cognitive Behavioural Therapy (CBT) for OCD — A brief 5-session CBT face-to-face intervention (therapist supported, involving workbooks) for adolescent Obsessive Compulsive Disorder (OCD). The brief CBT consists of 5 sessions of 60 to 90-minutes, with the option of 2 additional booster sessions (also 60 to 90 minutes), spanning a total of 24 weeks. The intervention includes home tasks, completion of regular routine outcome measures and participants listening to audio-recordings of the therapy sessions. The intervention sessions are delivered by routine child and adolescent mental health services (CAMHS) practitioners and take place in NHS and NHS-commissioned child and adolescent mental health services.

SUMMARY:
Obsessive-Compulsive Disorder (OCD) is a common and often disabling condition in young people, characterised by distressing, intrusive thoughts, images or urges, and repetitive behaviours intended to reduce discomfort or prevent harm. Around 1% of adolescents in the UK experience OCD, with many cases beginning in childhood or adolescence. Cognitive Behavioural Therapy (CBT) is the recommended treatment for OCD in young people, but access to treatment is limited due to high demand, long waiting lists, and lack of trained clinicians.

A brief form of CBT for OCD, supported by workbooks, has previously shown promising results in research settings. However, it remains unclear whether this approach is feasible, acceptable, and effective when delivered within routine NHS child and adolescent mental health services (CAMHS), especially for young people with co-occurring autism.

This single-arm feasibility trial aims to explore whether brief CBT can be delivered effectively in routine NHS and NHS-commissioned services to young people aged 11-18 years with OCD as their main presenting problem. The trial will also assess whether the intervention is acceptable to young people, their parents/carers, and clinicians, and whether outcomes are comparable to existing evidence.

Intervention Overview: The brief CBT intervention consists of five core sessions, with the option of two additional booster sessions, delivered over 24 weeks. Sessions are delivered face-to-face by trained clinicians and last between 60 to 90 minutes. The intervention is supported by a series of co-designed workbooks to be completed by the young person between sessions. Parents/carers are also provided with a workbook and encouraged to support the young person's progress where appropriate. Sessions may take place in the clinic or in other agreed settings, such as at home or school. The frequency of sessions decreases over time, with the first four sessions delivered weekly and later sessions spaced further apart.

The intervention includes psychoeducation, developing a cognitive-behavioural understanding of OCD, goal setting, and techniques to support motivation and engagement. A key focus is helping young people develop cognitive flexibility by testing and challenging unhelpful beliefs that drive OCD behaviours, supported by behavioural experiments. Parents/carers and other adults in the young person's life may also be involved to help generalise learning and promote progress.

Trial Aims: The trial has two primary aims:

To establish whether brief CBT for OCD can be delivered with fidelity and acceptability by clinicians in NHS services, and is acceptable to young people and their families.

To explore whether the intervention is associated with significant improvements in OCD symptoms for young people, including those with autism or high levels of autistic traits.

Trial Design: The study is a single-arm feasibility trial. Between 20-30 young people aged 11-18 years will be recruited alongside their parents/carers. Approximately 8-10 clinicians will be trained to deliver the intervention. OCD symptoms, treatment processes, and acceptability will be assessed at baseline, post-treatment (12 weeks), and at 3-month follow-up (24 weeks). Additional measures will be collected before each therapy session.

Qualitative interviews will be conducted with young people, parents/carers, and clinicians to understand their experiences of the intervention. Acceptability will also be measured using standardised questionnaires completed during and after treatment.

Outcomes: The primary outcomes are feasibility and acceptability of the intervention, assessed through session attendance, participant engagement, clinician adherence, and feedback from young people, parents/carers, and clinicians.

Secondary outcomes include changes in OCD symptoms, responsibility beliefs, family accommodation, and overall functioning, as well as measures of anxiety and depression. Data will be analysed to assess changes from baseline to post-treatment and follow-up, including for young people with and without autistic traits. Treatment adherence and clinician competence will also be evaluated.

DETAILED DESCRIPTION:
Background and Study Aims

Obsessive-Compulsive Disorder (OCD) is characterised by persistent, distressing intrusive thoughts, urges or images (i.e., intrusions) and behaviours aimed at preventing harm and reducing associated discomfort (e.g., compulsions or avoidance) (American Psychiatric Association, 2013). It affects around 1% of adolescents aged 11-19 years in the UK (Sadler et al., 2018), with up to 36% of OCD cases having an onset in adolescence across the globe (Dell'Osso et al., 2016).

The research team developed a brief 5 session CBT intervention (therapist supported, involving workbooks) for adolescent Obsessive Compulsive Disorder (OCD) which was evaluated through a large randomised control trial (RCT; Bolton et al., 2011, https://doi.org/10.1111/j.1469-7610.2011.02419.x) and found to be effective. In this trial, clinicians were all highly trained clinical psychologists and young people with 'marked symptoms of autistic spectrum disorder' were not included. The research team recently updated the materials (e.g., workbooks, treatment manual, training materials) with PPI and stakeholder involvement (https://doi.org/10.31234/osf.io/tcqm8).

This study aims to explore the feasibility of adopting brief CBT within NHS and NHS-commissioned child and adolescent mental health services. Specifically, we aim to ascertain whether brief CBT for adolescent OCD is:

1. Deliverable within services (i.e. whether clinicians show high levels of treatment adherence) and is acceptable to adolescents, their parents/carers and clinicians/service providers.
2. Associated with significant improvements in OCD symptoms and outcomes equivalent to outcomes for adolescent OCD within meta-analyses for all young people in the trial (including those with an autistic diagnosis and/or high levels of autistic traits).
3. Associated with significant improvements in OCD processes, functional interference, anxiety and depression symptoms.

   The researchers will examine this across the whole sample and those with an autism diagnosis and/or high levels of autistic traits.

   What does the study involve

   The brief CBT consists of 5 sessions of 60 to 90-minutes, with the option of 2 additional booster sessions (also 60 to 90 minutes), spanning a total of 24 weeks.

   Young people who meet diagnostic criteria for OCD via the Anxiety Disorders Interview Schedule for DSM-5 (ADIS-5) and all other inclusion criteria will be identified within the clinics, provided with written information about the study and invited to take part. Informed consent with be provided by young people aged 16 years or older. Young people under the age of 16 years will provide informed assent and their parent/carer will provide informed consent.

   Self-report questionnaire measures will be administered to young people and parents/carers at baseline (1-2 weeks prior to treatment), post-treatment (at 12 weeks) and 3-month follow-up (at 24 weeks). The CY-BOCS-II clinical interview will also be conducted with the young person and parent/carer at baseline and a 3-month follow-up.

   The young people receiving the treatment are expected to read and complete a total of six workbooks (an introduction workbook and five session-related workbooks) independently between sessions. As well as reading and completing the exercises in the workbooks, adolescents are also expected to complete tasks between sessions at home, or in the relevant context (e.g., school). Parents/carers may have some involvement in treatment sessions (depending on the preferences of the young person).

   The research team will also conduct qualitative interviews with young people and clinicians/service providers and administer a measure of treatment satisfaction to explore the acceptability of treatment. Depending on the preference of the participant, interviews will take place at the clinical site they are receiving treatment (young person) or they work for (clinician/service provider), at the University of Oxford, or online via MS Teams.

   What are the possible benefits and risks of participating?

   The young people who are participating will receive an evidence-based treatment for OCD. Brief CBT for adolescent OCD has potential benefits that they can use the skills taught and resources provided to them to continue to support a self-guided progress when faced with remaining symptoms or a relapse of symptoms. The clinicians delivering the treatment will be trained in a new treatment approach. This trial includes discussing potentially sensitive information with young people and parents/carers as part of the diagnostic interviews, intervention and self-report measures. Assessments will be conducted by trained assessors who have had DBS checks, have received extensive training to undertake assessments, and receive regular supervision from experienced clinicians within the research team. If any participant becomes distressed, assessors are trained to be able to handle this in a sensitive way and there will always be a named trained clinician from the research team available to speak to as part of a risk rota. In addition, the lead researchers for this study (PW and PS) are Consultant Clinical Psychologists experienced at recognising and managing potential distress.

   There will be a greater burden on all participants (young people, parents/carers and clinicians) than in routine clinical work in terms of their participation in assessment procedures. To minimise this burden, only measures that are strictly necessary are included. Clinician interviews will be carried out during the working day so that this does not create additional burden. Because qualitative interviews with young people are an additional time burden, they will be reimbursed for their time.

   When is the study starting and how long is it expected to run for?

   The study plans to run from 31/03/2025 to 31/03/2026.

   Recruitment

   All participants (young people, parents/carers, and clinicians) will be recruited from the Anxiety and Depression in Young People (AnDY) Research Clinics based in Oxford and Reading. The Oxford-based AnDY clinic is a collaboration with Oxford Health NHS Foundation Trust Child and Adolescent Mental Health Services (CAMHS). The Reading-based AnDY clinic is based in the School of Psychology and Clinical Language Sciences at the University of Reading and receives referrals through other local health and social care providers, including Berkshire Healthcare NHS Foundation Trust CAMHS. Both clinics provides assessment and brief psychological interventions to young people with anxiety disorders, depression or OCD and are informed by Children and Young People's Improving Access to Psychological Therapies (CYP IAPT) principles, enabling young people and their families to access high-quality, evidence-based treatments and research opportunities.

   Young people and their parents/carers who meet eligibility criteria for the study will be identified by the clinical team following their initial assessment. They will be approached and provided with participant information sheets. If they are interested in taking part, their details will be passed to the research team, and a member of the research team will speak to them in-person or by video call (via MS Teams) to answer questions and check understanding of the study. If they agree to take part, written informed consent will be obtained.

   Clinicians who meet eligibility criteria will be identified by the research team and trial site before the recruitment of young people with OCD. They will be approached and provided with participant information sheets. If they are interested in taking part, a member of the research team will speak to them in-person or by video call (via MS Teams) to answer questions and check understanding of the study. If they agree to take part, written informed consent will be obtained.

   Screening and Eligibility Assessment

   Eligibility for young people and their parent/carer to take part in the study is determined by the young person meeting criteria for a primary diagnosis of OCD, as assessed by the clinical team using the Anxiety Disorders Interview Schedule (ADIS-5-C/P; Silverman & Albano, 2024). The ADIS C/P is a structured interview to determine whether the young person meets diagnosis for OCD and/or a range of anxiety and behavioural disorders. Each diagnosis is given a corresponding clinician severity rating (CSR); the primary diagnosis is the disorder with the highest CSR. This assessment is part of the routine clinical service in both clinics. It is completed by a suitably trained assessor, under the clinical supervision of an experienced clinician and typically lasts three to four hours. The maximum duration allowed between a diagnostic assessment and registration in the trial is 6 months. Protocol waivers are not permitted; each participant must satisfy all the approved inclusion and exclusion criteria of the protocol. The clinical team will review the outcome of the diagnostic interview and other information to determine if the young person and parent/carer is eligible to take part.

   Eligibility for clinicians to take part in the study will be determined by evidence of adequate training, as outlined in the inclusion criteria.

   The research team will then review this information to confirm eligibility. This will be done anonymously (i.e., clinicians will not reveal names or any personally identifying information about the young person until informed consent for data sharing from young people (and parents, where applicable), has been obtained).

   Informed Consent

   Informed consent form will be provided to eligible participants by a suitably trained member of the clinical or research team. It will be provided no less than 24 hours after the participant has received study information, which is presented to the participant after eligibility to the trial has been determined (i.e., after the initial assessment and supervision).

   For young people and parent/carers, if they agree to participate in the trial, they both (regardless of age) must personally sign and date the latest approved version of the Informed Consent Form (or Assent Form for young people under 16 years of age) before any trial specific procedures are performed. This can be either the paper version, or the online version (worded the same as the paper version and administered via a secure online system such as Qualtrics). If consent is collected online, an appropriate electronic signature will be obtained (typing their full name). This will be done with a member of the research team (or a member of the clinical team acting on the behalf of the research team) either in person or on Microsoft Teams. As young people aged 16-18 years are providing their own informed consent, it will not be necessary for their parent/carer to be present. Signed informed consent will need to be obtained for any young people who turn 16 during participation within the study. A suitably trained member of the clinical or research team will share the Participant Information Sheet for 16-18 year olds and ask the young person to sign the Informed Consent Form prior to any further research activity.

   For clinicians, if they agree to participate, they must personally sign and date the latest approved version of the Informed Consent Form before completing any research activities. If consent is collected online, an appropriate electronic signature will be obtained (typing their full name).

   Written and verbal versions of the Participant Information Sheets and Informed Consent Forms will be presented to participants detailing the exact nature of the trial, what it will involve for the participant, the implications and constraints of the protocol, and any risks involved in taking part. For young people and parents/carers, it will be clearly stated that the participant is free to withdraw from the trial at any time for any reason without prejudice to future care. For all participants, it will be clear that they may withdraw without affecting their legal rights and with no obligation to give the reason for withdrawal.

   The participant will be allowed as much time as wished to consider the information, and the opportunity to question the Investigator, their GP and clinical team (where appropriate) or other independent parties to decide whether they will participate in the trial. Written Informed Consent will then be obtained by means of participant dated signature and dated signature of the person who presented and obtained the Informed Consent. The person who obtained the consent must be suitably qualified and experienced and have been authorised to do so by the Chief/Principal Investigator. A copy of the signed Informed Consent will be given to the participant. The original signed form will be retained at the trial site.

   Enrolment

   Young people and their parent/carer

   This trial does not include randomisation. Instead, if a young person is eligible, and agrees to take part in the study, the following procedure is in place. Once informed consent (or assent) is collected from both the young person and the parent/carer, the member of the clinical/research team assessing the young person will inform the Chief Investigator. They will also pass across demographic and baseline clinical information to the research team and the young person's GP will be informed by letter. The research team will then give the young person a unique research ID for the study. They will be placed on the treatment waiting list for treatment to start in the clinic with a suitably trained clinician as soon as possible.

   Clinicians

   If a clinician is eligible, agrees to take part and has provided written informed consent, the research team will allocate them a unique research ID for the study. Clinicians will then be able to be allocated to deliver the intervention to young people within the trial.

   Description of study procedure(s)

   We will collect routine clinical data gathered prior to and during study participation as well as data collected specifically for research purposes during the course of the research study. Standard outcome measures which are used in NHS care and assess OCD and related symptoms and processes will be administered throughout treatment, and at follow-ups. Self-report measures of OCD processes will be completed by the young person. These will typically be completed by young people and parents/carers at home and brought to the clinic. If they have difficulties completing measures, appropriate support will be provided by clinicians or members of the research team, as appropriate. Young people, parents/carers and clinicians will also complete measures related to treatment engagement and satisfaction. Diagnostic interviews using the will be conducted with the young person, and also with their parent/carer where possible at baseline (screening) as part of the routine clinical service. Therapists will also have regular review meetings with the research team, as well as sessions being video recorded to ensure treatment fidelity. In the participating services it is routine practice to video record therapy sessions to guide treatment and for supervision. Consent/assent will be sought from families for the use of the video or audio material of sessions for research purposes.

   The research team will also conduct qualitative interviews with the young people and clinicians/service providers and administer a measure of treatment satisfaction to explore the acceptability of treatment. For interviews with young people, demographic and clinical information will be used to inform sampling (i.e., to ensure that we recruit a maximum variation sample with respect to characteristics such as co-occurring mental health diagnoses and presence of autism/high level of autistic traits), and to provide context to the interview data. Semi-structured qualitative interviews lasting no more than one hour will be carried out with young people who received the treatment in the clinic or via video or telephone call. We will also interview clinicians at their place of work or via video or telephone call, asking about their experiences of delivering the treatment at the end of the study.

   Early Discontinuation/Withdrawal of Participants

   Participants in this study have the right to withdraw at any time and without providing a reason. Participants may also withdraw their consent, meaning that they wish to withdraw from the study completely. Should a participant choose to stop treatment and/or study assessments, all efforts will be made to report the reason for withdrawal as thoroughly as possible. Should a participant only wish to withdraw from therapy, efforts will be made to continue to obtain follow-up data with the permission of the participant. Participants can withdraw from the study, but any data obtained up until the point of withdrawal will be retained for use in the study analysis. No further data would be collected after withdrawal.

   After complete withdrawal, young people will continue with their routine NHS care. No follow-up observations will be required, but, as with therapy withdrawal, all attempts will be made to report the reason for withdrawal when participants inform the study team of their wish to withdraw.

   In addition, the Investigator may discontinue a participant from the trial treatment at any time if the Investigator considers it necessary for any reason including, but not limited to:

   Ineligibility (either arising during the trial or retrospectively having been overlooked at screening).

   The participant loses capacity to consent during the study. Significant protocol deviation. Significant non-compliance with treatment regimen or trial requirements. An adverse event which requires discontinuation of the trial intervention or results in inability to continue to comply with trial procedures.

   A significant increase in symptoms which requires discontinuation of the trial intervention or results in inability to continue to comply with trial procedures.

   A significant increase in risk to themselves or from others that cannot be managed by the current clinician.

   If the participant is withdrawn due to an adverse event, the Investigator will arrange for follow-up visits or telephone calls until the adverse event has been resolved or stabilised.

   If the withdrawing participant is a clinician and they are part-way through delivering the intervention to a young person, the young person will complete treatment with another clinician participating in the study. The number of withdrawals from treatment and/or follow-up measures will be logged with a summary of their reasons (if offered by the participant).

   Definition of End of Study

   The end of the study will be the date of the last point of data collection. This will be the last qualitative interview with the clinician participant. This will occur after all treatment sessions, follow-up measures and assessments and qualitative interviews with young people have been completed.

   Safety reporting

   Safety reporting will be in place in all instances taking place between the time a participant consents until the end of trial, as defined in the previous section. Follow up of any adverse events by the research team will take place up until the point that appropriate procedures are completed.

   Description of the Statistical Methods

   Analyses will investigate recruitment and retention rates presented as a CONSORT diagram providing results at all assessment points. Data completeness will be summarised for all clinical outcomes at each timepoint. Missing data will be explored to establish whether this is due to lack of response to specific questions, to the measure altogether or to loss of follow-up. All outcomes are continuous and will be summarised with means and standard deviations and minimum and maximum values. There will be no tests of statistical significance.

   For changes in OCD symptoms (on the CY-BOCS-II and OCI-CV-R), pre- to 24-week assessment effect sizes (Cohen's d) with 95% confidence intervals will be reported. For the CY-BOCS-II, we will also calculate treatment 'response' (>35% reduction in score and a Global Improvement score of 5 or 6) and 'remission' (a score ≤12 and Global Severity rating of 0, 1 or 2). We will also calculate pre- to 24-week assessment effect sizes (Cohen's d) with 95% confidence intervals for OCD process measures (CRIQ and CRAS), anxiety and depression symptoms (RCADS-C/P) and symptom interference (WSAS-Y-C/P). This will be done for the whole sample as well as those with and without an autism diagnosis and/or scoring above clinical cut-offs on a measure of autistic traits. Clinical outcomes will be examined to assess whether the observed effect sizes are in line with the expected effect based on those obtained in recent meta-analyses.

   We will also calculate reliable change for all clinical outcome and process measures (CY-BOCS-II, OCI-CV-R, CRIQ, CRAS, FAS-PR, RCADS-C/P, WSAS-Y-C/P) from pre- to 24-week assessment. Again, this will be done for the whole sample as well as those with and without an autism diagnosis and/or scoring above clinical cut-offs on a measure of autistic traits.

   Sample Size Determination

   As is typical in feasibility studies, the sample size is not based upon a power calculation (Arain et al., 2010). We aim to recruit 20 to 30 participants. If adverse events or significant deterioration were likely to occur as a result of participating in the trial, this would be expected to be observable within this sample size, and there will be sufficient throughput of potential participants within the recruitment period to examine recruitment and retention rates and participant flow through the trial and to examine fidelity of treatment (Julious, 2005; Lancaster et al., 2004; Sim & Lewis, 2012).

   A subsample will be involved in qualitative interviews after the treatment has been delivered. We will use purposive sampling and sample for a diverse range of demographic and clinical characteristics. The adequacy of the sample size will be continuously evaluated during the study, and recruitment to the interviews will come to an end when the sample holds sufficient information power to develop new knowledge (Braun & Clarke, 2019; Malterud et al., 2016). However, it may also be shaped and constrained by the number of potential interviewees, particularly in the clinician sample, as well as time and resources available.

   Who is funding the study?

   The funding is from an NIHR Applied Research Collaboration.

   Who is the main contact?

   The Chief Investigator is Dr. Polly Waite, polly.waite@psy.ox.ac.uk The study contact email address is ocd-yp@psy.ox.ac.uk

ELIGIBILITY:
Inclusion Criteria:

Young people:

* Willing and able to give informed assent (if aged 11-15 years, and parent/carer consent is provided) or consent (if aged 16-18 years) for participation in the study.
* Aged 11 to 18 years at the time of recruitment.
* Diagnosed with OCD using the Anxiety Disorders Interview Schedule (ADIS) and OCD has been identified as the primary problem.
* If on pharmacotherapy for OCD, then stable dose for at least 6 weeks prior to trial entry.
* Able to speak and read English at a sufficient level to be able to read and understand the workbooks and materials and complete exercises in the workbooks.
* Willing to engage in the treatment.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Parents/carers:

* Able and willing to provide written informed consent for their child's participation in the study.
* Able to read the parent/carer workbook and materials.
* Willing and able to participate.

Clinicians:

* Working within a participating NHS or NHS-commissioned service.
* Have a professional qualification in psychological therapy that includes training in CBT at or above post-graduate certificate level.
* Willing to participate.
* Clinical capacity and managerial approval to participate

Exclusion Criteria:

Young people:

* The clinical assessment indicates that risk/safeguarding cannot be safely managed within the service.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Evidence of learning difficulties identified by schools or evident at interview that would inhibit participation in cognitive components of therapy.
* Currently receiving a psychological intervention for OCD.

Parents/carers:

* No exclusion criteria.

Clinicians:

* No exclusion criteria

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Credibility and Expectation of Treatment Questionnaire (CEQ; Borkovec & Nau, 1972) | Baseline and follow-up (week 24)
  The Credibility and Expectation of Treatment Questionnaire (CEQ; Borkovec & Nau, 1972) will be collected at baseline and used to establish treatment acceptability. Score range 0-30. Higher scores represent a better outcome.
Experience of Service Questionnaire (ESQ; Astride-Stirling, 2002) | End of treatment (week 12) and follow-up (week 24)
  The Experience of Service Questionnaire (ESQ; Astride-Stirling, 2002) will be used at the end of treatment (Week 12) and follow-up (Week 24) to measure young peoples' and parent/carers' expectations and views on the acceptability of the treatment and service.
Therapist Experience of Training and Treatment Delivery Questionnaire | Follow-up (week 24)
  The Therapist Experience of Training and Treatment Delivery Questionnaire will be given to clinicians at follow-up (Week 24) in order to establish their perceived competence, acceptability and feasibility in delivering the intervention. Score range 19-95. Higher scores represent a better outcome.
Attrition Rate | From enrolment to the end of follow-up (week 24)
  Feasibility will also be established by the number and rate of participants who drop-out of treatment (attrition rate).
Therapist Adherence | From enrolment to the end of treatment (week 12)
  Recordings of therapy sessions will be rated by the research team to assess therapist competency and intervention adherence.
Semi-structured interviews | At follow-up (week 24)
  Semi-structured one-to-one/joint interviews at follow-up (Week 24) exploring experiences of receiving/delivering the treatment will be conducted with participants (young people and clinicians).
Participant Engagement with Materials | From first intervention session (week 1) to the end of treatment (week 12)
  A brief questionnaire for clinicians to rate whether the workbooks were not completed, partially completed or fully completed by the young person. To be completed following each clinical session with workbooks.
Session Rating Scale (SRS; Miller, Duncan & Johnson, 2002) | From first intervention session (week 1) to the end of follow-up (week 24)
  The Session Rating Scale is a brief, four-item measure developed to assess the therapeutic alliance from the client's perspective in real-time. Higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Children's Yale-Brown Obsessive Compulsive Scale II (CY-BOCS-II; Abramovitch et al., 2022) | Baseline and follow-up (week 24)
  The Children's Yale-Brown Obsessive Compulsive Scale II (CY-BOCS-II; Abramovitch et al., 2022), the gold-standard in the assessment of the symptoms and severity of OCD in young people (Rapp et al., 2016) will be used at baseline and at follow-up (Week 24). The CY-BOCS-II will be used to measure change in OCD severity. Score range 0-50. Lower scores represent a better outcome.
Obsessive-Compulsive Inventory - Child Version - Revised (OCI-CV-R; Abramovitch et al., 2022) | From baseline to follow-up (week 24)
  The Obsessive-Compulsive Inventory - Child Version - Revised (OCI-CV-R; Abramovitch et al., 2022) is a self-report measure of OCD symptoms and will be collected at baseline and every subsequent contact with the young people (each clinical session, post-intervention at Week 12 and follow-up at Week 24). Score range 0-36. Lower scores represent a better outcome.
Child Responsibility Interpretations Questionnaire - CRIQ (Salkovskis & Williams, 2004a; Salkovskis & Williams, 2004b) | From baseline to follow-up (week 24)
  A measure of the OCD maintenance processes of responsibility beliefs will be collected at baseline and each clinical session to measure process changes and inform clinical treatment (Salkovskis & Williams, 2004a; Salkovskis & Williams, 2004b).
Child Responsibility Attitude Scale - CRAS (Salkovskis & Williams, 2004a; Salkovskis & Williams, 2004b) | From baseline to follow-up (week 24)
  A measure of the OCD maintenance processes of responsibility attitudes will be collected at baseline and each clinical session to measure process changes and inform clinical treatment (Salkovskis & Williams, 2004a; Salkovskis & Williams, 2004b).
Family Accommodation Scale-Parent Report (FAS-PR) (Peris et al., 2008; Storch et al., 2007) | Baseline, end of treatment (week 12) and at follow-up (week 24).
  The Family Accommodation Scale-Parent Report (FAS-PR) (Peris et al., 2008; Storch et al., 2007) will also be completed by parent/carers in order to assess family members' participation in or facilitation of the young person's OCD-related behaviours. Score range 0-36. Lower scores represent a better outcome.
Demographic information | Baseline
  As part of normal clinical practice, additional baseline data will be collected, including demographic information (including age, gender, ethnicity, parental education and occupation) and clinical information (including diagnostic and self-report questionnaire data and use of medication).
Autism-Spectrum Quotient-Short (AQ-Short; Hoekstra et al., 2011) | Baseline
  At baseline we will also collect a measure of autistic traits from the Autism-Spectrum Quotient-Short (AQ-Short; Hoekstra et al., 2011)
Work and Social Adjustment Scale - Youth version (WSAS-Y; Jassi et al., 2020) | Baseline, post-intervention (week 12) and follow up (week 24)
  A measure of functional interference of the OCD (WSAS-Y; Jassi et al., 2020). Score range 0-40. Lower scores represent a better outcome.
Revised Child Anxiety and Depression Scale (RCADS; Chorpita et al., 2000) | From baseline to follow-up (week 24)
  A routine measure of symptoms of anxiety and depression, the Revised Child Anxiety and Depression Scale (RCADS; Chorpita et al., 2000), will be completed by the young person and collected at each clinical session. Score range 0-141. Lower scores represent a better outcome.
Vancouver Obsessive Compulsive Inventory - Mental Contamination (VOCI-MC; Radomsky, Rachman, Shafran, Coughtrey, & Barber, 2014) | Baseline and follow-up (week 24)
  A 20-item self-report measure for mental contamination features of OCD. This measure will have a small adaptation to one question wording following Public-Patient Involvement. Lower scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - AnDY Research Clinic, Reading, Berkshire
  - Department of Experimental Psychology, Oxford, Oxfordshire
  - AnDY Research Clinic Oxford, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
After publication of results, the datasets will be de-identified and archived on a suitable data repository. The specific data repository is unknown and will be made available at a later date.
  Intention to publish date 01/06/2026

REFERENCES:
- [Background] Dell'Osso B, Benatti B, Hollander E, Fineberg N, Stein DJ, Lochner C, Nicolini H, Lanzagorta N, Palazzo C, Altamura AC, Marazziti D, Pallanti S, Van Ameringen M, Karamustafalioglu O, Drummond LM, Hranov L, Figee M, Grant JE, Zohar J, Denys D, Menchon JM. Childhood, adolescent and adult age at onset and related clinical correlates in obsessive-compulsive disorder: a report from the International College of Obsessive-Compulsive Spectrum Disorders (ICOCS). Int J Psychiatry Clin Pract. 2016 Nov;20(4):210-7. doi: 10.1080/13651501.2016.1207087. Epub 2016 Jul 19. PMID 27433835
- [Background] Bolton D, Williams T, Perrin S, Atkinson L, Gallop C, Waite P, Salkovskis P. Randomized controlled trial of full and brief cognitive-behaviour therapy and wait-list for paediatric obsessive-compulsive disorder. J Child Psychol Psychiatry. 2011 Dec;52(12):1269-78. doi: 10.1111/j.1469-7610.2011.02419.x. Epub 2011 Jun 3. PMID 21644984